CLINICAL TRIAL: NCT01490840
Title: A 6-month, Multicenter, Randomized, Controlled Parallel Group Study to Evaluate the Effect of Physical Training on Fatigue in Patients With Relapsing-remitting Multiple Sclerosis Treated With Fingolimod, Followed by a 6 Month Optional Extension Phase
Brief Title: Effect of Physical ACtivity in Fingolimod Treated patiEnts (PACE) With Relapsing-remitting Multiple Sclerosis
Acronym: PACE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study stopped due to slow enrollment and low participant compliance.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFTY720DDE07; 2011-002969-38 (EudraCT Number)
Record Dates: First submitted 2011-12-09; First posted 2011-12-13 (Estimated); Results first posted 2016-05-12 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-04

CONDITIONS: Fatigue in Multiple Sclerosis
Keywords: Fatigue; MS; Multiple Sclerosis; Exercise; Physical activity; Physical training; Fingolimod
MeSH Terms: conditions — Fatigue; Multiple Sclerosis; Motor Activity | interventions — Exercise

ARMS (2):
- E-training (Experimental): Fingolimod as baseline immunomodulatory multiple sclerosis treatment was prescribed as per clinical practice. During phase 1, participants randomized to this arm had an introductory group session, hosted by a sports therapist. The individual training schedule was comprised of strength exercises twice a week for 30-45 minutes and endurance training once a week for 20-60 minutes for 6 months. The participants documented each training session thoroughly via the web-based application (duration, type of exercises, number of repetitions and sets, perceived exertion). A standard course of corticosteroids (methylprednisolone) on an inpatient or outpatient basis was allowed for treatment of relapses as clinically warranted. Steroid treatment consisted of 3-5 days and up to 1,000 mg methylprednisolone/day. After 6 months, Phase 2, the same Phase 1 regimen applied.
  Interventions: Other: Physical exercise
- Waiting (Experimental): Fingolimod as baseline immunomodulatory multiple sclerosis treatment is prescribed as per clinical practice. During Phase 1, participants randomized to this arm did not receive e-training exercise. After a 6 months waiting period, phase 2, participants had an introductory group session, hosted by a sports therapist. The individual training schedule was comprised of strength exercises twice a week for 30-45 minutes and endurance training once a week for 20-60 minutes for 6 months. The participants documented each training session thoroughly via the web-based application (duration, type of exercises, number of repetitions and sets, perceived exertion). A standard course of corticosteroids (methylprednisolone) on an inpatient or outpatient basis was allowed for treatment of relapses as clinically warranted. Steroid treatment consisted of 3-5 days and up to 1,000 mg methylprednisolone/day.
  Interventions: Other: Physical exercise

INTERVENTIONS:
Other: Physical exercise — Strength training exercises are performed against own body weight or with training aids like elastic rubber bands or gym balls. All exercises are home-based. To increase balance and core stability, a subset of exercises is performed on shaky ground and/or one-legged. Exercise intensity, duration and frequency are individually assigned by a sports therapist. For each muscle group, a set of exercises of increasing difficulty allows for individual and progressive training adaption. Therapists can choose from an exercise database of approximately 150 different strength exercises with different graduation.

SUMMARY:
This study evaluated the effect of an individualized web-based physical training in fingolimod -treated patients.

DETAILED DESCRIPTION:
In this study, it was planned to randomize 226 participants. However, only 178 participants were randomized during a timeframe of 2 years and 8 months. Therefore, the study was terminated due to slow enrollment and low participant compliance to the physical training schedule.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with relapsing remitting MS defined by 2010 revised McDonald criteria
* Patients with Expanded Disability Status Scale (EDSS) score of 0-3.5 (including)
* Immunomodulatory treatment with prescribed fingolimod for at least one month prior to baseline
* Fatigue score assessed by mFIS of equal or greater than 14 at screening
* Neurologically stable with no evidence of relapse within 30 days prior to inclusion date

Exclusion Criteria:

* Patients who have been treated with:

  * systemic corticosteroids or immunoglobulins within 1 month prior to randomization;
  * immunosuppressive medications such as azathioprine, cyclophosphamide, or methotrexate within 3 months prior to randomization;
  * monoclonal antibodies (including natalizumab) within 3 months prior to randomization;
  * mitoxantrone within 6 months prior to randomization
  * cladribine at any time.
* Patients with any medically unstable condition, as assessed by the primary treating physician at each site.
* Patients with any of the following cardiovascular conditions :

  * history of cardiac arrest;
  * history of myocardial infarction or with current unstable ischemic heart disease;
  * history of angina pectoris due to coronary spasm or history of Raynaud syndrome
  * Heart failure (NYHA III-IV) or any severe cardiac disease as determined by the investigator;
  * history or presence of a second-degree AV block, Type II or a third-degree AV
  * block
  * patients receiving Class Ia (ajmaline, disopyramide, procainamide, quinidine) or
  * III antiarrhythmic drugs (e.g., amiodarone, bretylium, sotalol, ibulitide, azimilide,
  * dofelitide);
  * proven history of sick sinus syndrome or sino-atrial heart block;
  * uncontrolled hypertension
* Clinically relevant internal disease (e.g. uncorrected anemia) or orthopedic diseases (e.g. scoliosis) that might interfere with physical training
* Any severe disability or clinical impairment that can prevent the patient to meet all study requirements at the investigator's discretion

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2011-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (27):
- Germany (27):
  - Novartis Investigative Site, Dortmund, Germany
  - Novartis Investigative Site, Leipzig, Germany
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Alzenau in Unterfranken
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Bad Mergentheim
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Böblingen
  - Novartis Investigative Site, Erbach im Odenwald
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Prien am Chiemsee
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Sinsheim
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Teupitz
  - Novartis Investigative Site, Unterhaching

REFERENCES:
- [Derived] Maurer M, Schuh K, Seibert S, Baier M, Hentschke C, Streber R, Tallner A, Pfeifer K. A randomized study to evaluate the effect of exercise on fatigue in people with relapsing-remitting multiple sclerosis treated with fingolimod. Mult Scler J Exp Transl Clin. 2018 Feb 14;4(1):2055217318756688. doi: 10.1177/2055217318756688. eCollection 2018 Jan-Mar. PMID 29479457

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized1:1 to receive a structured physical intervention (e-training) or no physical intervention (waiting).
Pre-assignment Details: At the end of the 6 month core phase (phase 1), participants in the waiting group had the option to receive e-training for 6 months in the phase 2 optional extension. Participants in the e-training group had the option to continue their e-training for another 6 months in the phase 2 extension.
Groups:
- Waiting: Fingolimod as baseline immunomodulatory multiple sclerosis treatment is prescribed as per clinical practice. During Phase 1, participants randomized to this arm did not receive e-training exercise. After a 6 month waiting period, phase 2, participants had an introductory group session, hosted by a sports therapist. The individual training schedule was comprised of strength exercises twice a week for 30-45 minutes and endurance training once a week for 20-60 minutes for 6 months. The participants documented each training session thoroughly via the web-based application (duration, type of exercises, number of repetitions and sets, perceived exertion). A standard course of corticosteroids (methylprednisolone) on an inpatient or outpatient basis was allowed for treatment of relapses as clinically warranted. Steroid treatment consisted of 3-5 days and up to 1,000 mg methylprednisolone/day.
Period: Phase 1
Arm/Group | E-training | Waiting
Started | 94 | 84
Modified Full Analysis Set | 56 | 83
Completed | 84 | 78
Not Completed | 10 | 6
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Visit 6a omitted | 1 | 0
Period: Phase 2
Arm/Group | E-training | Waiting
Started | 81 (3 participants discontinued between phase 1 and phase 2) | 74 (4 participants discontinued between phase 1 and phase 2)
Completed | 75 | 68
Not Completed | 6 | 6
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Permanent interruption of fingolimod | 0 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | E-training | Waiting | Total
Number analyzed (Participants) | 94 | 84 | 178
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.9 (10.4) | 39.4 (8.7) | 40.2 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 57 | 122
  Male | 29 | 27 | 56

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Fatigue as Measured by the Modified Fatigue Impact Scale (mFIS ).
Description: The mFIS provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning. It is a 21-item, structured, self-report questionnaire that generally can be completed with little or no intervention from an interviewer. The mFIS score ranged from 0 (not tired) to 84 (tired). A negative change from baseline indicates improvement.
Time Frame: Baseline, 6 months
Population: Modified Full Analysis Set (ModFAS): The ModFAS included participants with sufficient e-training compliance.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | E-training | Waiting
Number analyzed (Participants) | 56 | 83
score on a scale | -3.57 (11.3) [-6.81 to -0.34] | -2.10 (12.1) [-4.69 to 0.49]
Statistical Analysis 1: Comparison: E-training vs Waiting; Test type: Non-Inferiority or Equivalence — A sample size of 90 in each group would have 80% power to detect a difference in means of 3.8, assuming that the common standard deviation is 9.05, using a two group t-test with a 0.05 2-sided significance level; p = 0.4579, ANCOVA; Mean Difference (Net) = -1.47, 95% CI 2-sided [-5.39 to 2.44]

2. Secondary Outcome: Change From Baseline in Isometric and Dynamic Muscular Strength as Measured by Sit-to-stand Test
Description: The Sit to Stand Test is a functional outcome measure of the lower-extremity muscle power. The test was performed 3 times with one minute rest in between. The best attempt out of three was used for the analysis. A positive change from baseline indicates improvement.
Time Frame: baseline, 6 months
Population: The ModFAS, which included participants with sufficient e-training compliance, was considered for the analysis. Only participants with both baseline and month 6 values were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: watt/kilogram body weight
Arm/Group | E-training | Waiting
Number analyzed (Participants) | 55 | 83
watt/kilogram body weight | 0.03 [-0.31 to 0.36] | 0.27 [-0.01 to 0.55]

3. Secondary Outcome: Change From Baseline in Isometric and Dynamic Muscular Strength as Measured by Change in Leg Strength and Trunk Strength
Description: Isometric and dynamic muscular strength was measured by an Isomed 2000 isometric measurement device (knee flexion/tension, trunk flexion/extension).
  Isomed 2000 device measures muscular flexion and tension under standardized training conditions. A positive change from baseline indicates improvement.
Time Frame: baseline, 6 months
Population: Modified Full Analysis Set (ModFAS): The ModFAS included participants with sufficient e-training compliance.
Measure: Least Squares Mean (95% Confidence Interval); unit: newton meter
Arm/Group | E-training | Waiting
Number analyzed (Participants) | 56 | 83
newton meter
  Leg strength | 0.50 [-1.83 to 2.83] | 1.63 [-0.32 to 3.58]
  Trunk strength | 0.08 [-0.01 to 0.18] | 0.12 [0.04 to 0.20]

4. Secondary Outcome: Change From Baseline in Isometric and Dynamic Muscular Strength as Measured by Leg Strength Endurance
Description: as for outcome 3
Time Frame: baseline, 6 months
Population: Modified Full Analysis Set (ModFAS): The ModFAS included participants with sufficient e-training compliance.
Measure: Least Squares Mean (95% Confidence Interval); unit: joule
Arm/Group | E-training | Waiting
Number analyzed (Participants) | 56 | 83
joule | 51.28 [-50.7 to 153.3] | 130.80 [47.53 to 214.1]

5. Secondary Outcome: Change From Baseline in Quality of Life as Measured by the Hamburg Quality of Life Questionnaire in Multiple Sclerosis (HAQUAMS)
Description: The Hamburg Quality of Life Questionnaire in Multiple Sclerosis (HAQUAMS) consists of 44 items, 28 of which are the basis for computation of five subscale scores reflecting major dimensions of health-related quality of life (HRQoL) in MS: Fatigue/Thinking (4 items), Mobility lower limb (5 items), Mobility upper limb (5 items), Social function (6 items) and Mood (eight items). Subscales and total score range from 1 to 5, with high scores indicating a lower quality of life. In this study, the total score and following 3 subscales: fatigue/thinking, mobility lower limb and mobility upper limb only were analyzed. A negative change from baseline indicates improvement.
Time Frame: Baseline, 6 months, 12 months
Population: Modified Full Analysis Set (ModFAS): The ModFAS included participants with sufficient e-training compliance.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | E-training | Waiting
Number analyzed (Participants) | 56 | 83
score on a scale
  Total score | -0.11 [-0.21 to -0.01] | -0.02 [-0.10 to 0.06]
  Fatigue/thinking | -0.30 [-0.48 to -0.12] | -0.16 [-0.30 to -0.01]
  Mobility lower limb | -0.00 [-0.16 to 0.15] | 0.08 [-0.04 to 0.20]
  Mobility upper limb | -0.00 [-0.10 to 0.10] | 0.12 [0.04 to 0.20]

6. Secondary Outcome: Change From Baseline in Fatigue as Measured by the WEIMuS (Würzburg Fatigue Inventory for MS)
Description: The WEIMuS (Würzburg Fatigue Inventory for MS) scale is a validated self-assessment instrument to quantify the degree of fatigue. The scale consists of 17 items with 5 categories that are scored from '0' to '4'. The subscores for cognitive and physical fatigue range from 0 to 36 and from 0 to 32, respectively, with the total sum score ranging from 0 to 68; higher scores indicate higher degrees of fatigue. A negative change from baseline indicates improvement.
Time Frame: Baseline, 6 months
Population: Modified Full Analysis Set (ModFAS): The ModFAS included participants with sufficient e-training compliance.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | E-training | Waiting
Number analyzed (Participants) | 56 | 83
score on a scale | -1.90 [-4.91 to 1.11] | -1.12 [-3.55 to 1.31]

7. Secondary Outcome: Change From Baseline in Depression as Measured by the Beck Depression Inventory Second Edition (BDI-II)
Description: The Beck Depression Inventory Second Edition (BDI-II) is a 21-item self-report instrument intended to assess the existence and severity of symptoms of depression as listed in the American Psychiatric Association's Diagnostic and Statistical Manual of Mental Disorders Fourth Edition. Each of the 21 items corresponding to a symptom of depression is summed to give a single score for the BDI-II. There is a four-point scale for each item ranging from 0 to 3. The total score ranges from 0 - 63. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe. A negative change from baseline indicates improvement.
Time Frame: Baseline, 6 months
Population: Modified Full Analysis Set (ModFAS): The ModFAS included participants with sufficient e-training compliance.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | E-training | Waiting
Number analyzed (Participants) | 56 | 83
score on a scale | -2.62 [-4.42 to -0.81] | -1.97 [-3.43 to -0.52]

8. Secondary Outcome: Change From Baseline in Aerobic Capacity (VO2max) as Measured by a Physical Endurance Spiroergometry on a Treadmill
Description: Physical endurance spiroergometry was accomplished. Ergometry was assessed according to national guidelines of the German society for sports medicine. Ergometry is a combined examination of circulation and lung function and was performed as a submaximal or maximal test depending on the participant's individual performance. A negative change from baseline indicates improvement.
Time Frame: Baseline, 6 months
Population: Modified Full Analysis Set (ModFAS): The ModFAS included participants with sufficient e-training compliance.
Measure: Least Squares Mean (95% Confidence Interval); unit: [ml/min/kg][watt/kg body weight]
Arm/Group | E-training | Waiting
Number analyzed (Participants) | 56 | 83
[ml/min/kg][watt/kg body weight] | -0.52 [-1.60 to 0.56] | -0.79 [-1.66 to 0.08]

9. Secondary Outcome: Change From Baseline in Peak Expiratory Flow as Measured by a Physical Endurance Spiroergometry on a Treadmill
Description: Physical endurance spiroergometry was accomplished. Ergometry was assessed according to national guidelines of the German society for sports medicine. Ergometry is a combined examination of circulation and lung function and was performed as a submaximal or maximal test depending on the participant's individual performance. A positive change from baseline indicates improvement.
Time Frame: Baseline, 6 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: L/s
Arm/Group | E-training | Waiting
Number analyzed (Participants) | 46 | 78
L/s | 0.05 [-0.15 to 0.24] | 0.01 [-0.15 to 0.17]

ADVERSE EVENTS:
Arm/Group | E-training | Waiting
Serious Adverse Events (participants affected / at risk) | 5/94 | 9/84
Other Adverse Events (participants affected / at risk) | 58/94 | 59/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E-training (N=94) | Waiting (N=84)
ARRHYTHMIA (Cardiac disorders) | 0 | 1
EXTRASYSTOLES (Cardiac disorders) | 0 | 1
PALPITATIONS (Cardiac disorders) | 0 | 1
APPENDICITIS PERFORATED (Infections and infestations) | 0 | 1
CONJUNCTIVITIS (Infections and infestations) | 0 | 1
BONE CONTUSION (Injury, poisoning and procedural complications) | 0 | 1
CONCUSSION (Injury, poisoning and procedural complications) | 0 | 1
DISLOCATION OF VERTEBRA (Injury, poisoning and procedural complications) | 1 | 0
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 0
ASTROCYTOMA, LOW GRADE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
EPILEPSY (Nervous system disorders) | 1 | 0
GENERALISED TONIC-CLONIC SEIZURE (Nervous system disorders) | 0 | 1
HEMIPARESIS (Nervous system disorders) | 1 | 0
ISCHAEMIC CEREBRAL INFARCTION (Nervous system disorders) | 1 | 0
MUSCLE SPASTICITY (Nervous system disorders) | 1 | 0
MENORRHAGIA (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | E-training (N=94) | Waiting (N=84)
DIARRHOEA (Gastrointestinal disorders) | 5 | 2
BRONCHITIS (Infections and infestations) | 3 | 8
NASOPHARYNGITIS (Infections and infestations) | 34 | 33
ORAL HERPES (Infections and infestations) | 6 | 2
SINUSITIS (Infections and infestations) | 5 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 5
BLOOD CHOLESTEROL INCREASED (Investigations) | 2 | 5
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 | 5
HEADACHE (Nervous system disorders) | 4 | 6
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 22 | 15
DEPRESSION (Psychiatric disorders) | 4 | 8
SLEEP DISORDER (Psychiatric disorders) | 10 | 4
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 8
HYPERTENSION (Vascular disorders) | 4 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.